CLINICAL TRIAL: NCT00006289
Title: Neurotropin for Acute Dental Pain and for Chronic Neuropathic Pain
Brief Title: Neurotropin to Treat Chronic Neuropathic Pain
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: difficulty in the recruitment of patients
Sponsor: National Institute of Nursing Research (NINR) (NIH)
Collaborators: National Institutes of Health Clinical Center (CC) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 000200; 00-NR-0200 (Other: NIH)
Record Dates: First submitted 2000-09-21; First posted 2000-09-22 (Estimated); Results first posted 2016-06-21 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Complex Regional Pain Syndrome Type I; Complex Regional Pain Syndrome Type II
Keywords: Analgesia; Causalgia; CRPS; Neuropathic Pain; Oral Surgery; Reflex Sympathetic Dystrophy; Sympathetic Nervous System; Chronic Regional Pain Syndrome
MeSH Terms: conditions — Complex Regional Pain Syndromes; Causalgia; Agnosia; Neuralgia; Reflex Sympathetic Dystrophy | interventions — neurotropin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo first, then Neurotropin (G-1) (Active Comparator): Double blind cross-over study: receive placebo for 5 weeks and then Neurotropin for 5 weeks (after at least 1 week washout period). Assignment to each group was in random order, selected by the pharmacy with all others blind.
  Interventions: Drug: Placebo; Drug: Neurotropin
- Neurotropin first, then Placebo (G-2) (Active Comparator): Double blind cross-over study: receive Neurotropin for 5 weeks and then placebo for 5 weeks (after at least 1 week washout period). Assignment to each group was in random order, selected by the pharmacy with all others blind.
  Interventions: Drug: Placebo; Drug: Neurotropin

INTERVENTIONS:
Drug: Placebo — 4 tabs b.i.d.
  Other Names: Drug A
Drug: Neurotropin — 4 tabs b.i.d.
  Other Names: Drug B

SUMMARY:
This study will examine the effectiveness of the drug neurotropin in treating chronic pain after injury to a limb or a large nerve.

Two groups of patients will participate in this study: patients with complex regional pain syndrome type 1, or CRPS-I (also called reflex sympathetic dystrophy) and patients with complex regional pain syndrome type 2, or CRPS-II. CRPS-I is pain that develops after relatively minor injury to an arm or leg, but lasts much longer and is much more severe than would normally be expected. CRPS-II is pain resulting from injury to a large nerve. Candidates will have a history and physical examination, blood tests, and electrocardiogram. Participants will undergo the following tests and procedures:

Patients with CRPS I and II will receive an individualized regimen of physical therapy and standard treatment to control their pain. In addition, they will receive neurotropin or placebo tablets for 5 weeks, then no trial medicine for at least 1 week, and then the other trial drug for the next 5 weeks. That is, patients who took placebo the first 5 weeks will take neurotropin the second 5 weeks and vice versa. Neither the patients nor the doctors will know who received which drug during the two intervals until the study is over. Patients will complete questionnaires about their pain, quality of life, and ability to perform daily living activities. They will have various tests to measure pain (such as sensitivity to heat and cold, to an electric current, to a mild pin prick, etc.); to provide information about changes in their condition (such as tests of range of motion of joints and limb size); to measure blood circulation and sweating in the arm or leg (such as measurements of blood flow to the limb, skin temperature, and sweat production), and other procedures.

DETAILED DESCRIPTION:
Patients with Reflex Sympathetic Dystrophy (RSD), re-named Complex Regional Pain Syndrome, type I (CRPS-I), have chronic, post-traumatic pain that spreads beyond the distribution of any single peripheral nerve without evidence of major peripheral nerve damage. A similar disorder, Causalgia, re-named CRPS-II, presents with clear evidence of nerve injury. No successful drug treatment exists for these disorders. Neurotropin is a non-protein extract of cutaneous tissue from rabbits inoculated with vaccinia virus. Neurotropin has been used extensively in Japan to treat RSD and other painful conditions; however, the drug has not undergone clinical therapeutic testing in the United States. This protocol is to carry out double-blind, placebo-controlled, crossover studies about clinical efficacy of Neurotropin for acute pain in dental outpatients and for chronic pain in outpatients with CRPS-I or II.

ELIGIBILITY:
* INCLUSION CRITERIA:

CRPS patients are referred with a diagnosis of CRPS-I or CRPS-II in one limb only, based on pain (1) that is post-traumatic and spread beyond the region of the injury; (2) has persisted for more than 2 weeks; and (3) is associated with swelling, altered skin color or skin temperature, altered sweating, allodynia or hyperesthesia or limitation of active movement. Atrophic changes in skin, hair loss or nail changes, or disuse atrophy of skeletal muscle may be present.

Both sexes are to be studied.

All ethnic and racial groups can participate.

Patients must be willing to return to NIH for follow-up evaluation under this protocol.

EXCLUSION CRITERIA:

Pregnant and lactating women are excluded.

Based on the oral surgeon's postoperative diagnosis, any extraction which is classified as producing unusual surgical trauma will result in exclusion from the remainder of the study.

Dental subjects will also be excluded if they are not adequately sedated by midazolam alone and require intraoperative administration of an opioid drug such as fentanyl, administration of greater than 14.4 ml of local anesthetic (2% lidocaine with 1:100,000 epinephrine), or postoperative administration of a steroid for possible injury to the inferior alveolar nerve.

Patients referred with CRPS-I or CRPS II who have abnormal screening test results or who have non-traumatic disorders to which pain may be attributed (gout, malignancy, arthritis, etc.) will be excluded.

Any patients who have had ablative procedures for treatment of their neuropathic pain disorder will not be eligible for inclusion in this study.

Patients who have a positive HIV result will be excluded.

Subjects with obviously impaired mental capacity that precludes informed consent and ability to provide adequate self-ratings are to be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2000-09; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leorey Saligan, PhD, CRNP, Principal Investigator — National Institute of Nursing Research (NINR)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Stanton-Hicks M, Janig W, Hassenbusch S, Haddox JD, Boas R, Wilson P. Reflex sympathetic dystrophy: changing concepts and taxonomy. Pain. 1995 Oct;63(1):127-133. doi: 10.1016/0304-3959(95)00110-E. PMID 8577483
- [Background] Galer BS, Bruehl S, Harden RN. IASP diagnostic criteria for complex regional pain syndrome: a preliminary empirical validation study. International Association for the Study of Pain. Clin J Pain. 1998 Mar;14(1):48-54. doi: 10.1097/00002508-199803000-00007. PMID 9535313
- [Background] Bruehl S, Harden RN, Galer BS, Saltz S, Bertram M, Backonja M, Gayles R, Rudin N, Bhugra MK, Stanton-Hicks M. External validation of IASP diagnostic criteria for Complex Regional Pain Syndrome and proposed research diagnostic criteria. International Association for the Study of Pain. Pain. 1999 May;81(1-2):147-54. doi: 10.1016/s0304-3959(99)00011-1. PMID 10353502

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Most patients are recruited by direct physician referral or through the Patient Recruitment and Public Liaison (PRPL) office. Potential subjects are determined to be qualified by screening at Clinical Center, NIH in the US.
Pre-assignment Details: Patients who have abnormal results from routine laboratory test or are positive for HIV are excluded. Women who are pregnant or positive for pregnancy test are excluded. Also patients who have non-traumatic pain disorders or are obviously have impaired mental capacity are excluded.
Groups:
- Placebo First, Then Neurotropin: Receive the placebo b.i.d. for 5 weeks and then Neurotropin b.i.d. for 5 weeks (after at least 1 week washout period)
- Neurotropin First, Then Placebo: Receive Neurotropin b.i.d. for 5 weeks and then the placebo b.i.d. for 5 weeks (after at least 1 week washout period)
Period: First Intervention (5 Weeks)
Arm/Group | Placebo First, Then Neurotropin | Neurotropin First, Then Placebo
Started | 11 | 10
Completed | 10 | 10
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Washout (>= 1 Week)
Arm/Group | Placebo First, Then Neurotropin | Neurotropin First, Then Placebo
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Second Intervention (5 Weeks)
Arm/Group | Placebo First, Then Neurotropin | Neurotropin First, Then Placebo
Started | 10 | 10
Completed | 9 | 9
Not Completed | 1 | 1
Not completed — Protocol Violation | 1 | 1

BASELINE CHARACTERISTICS:
Population: Clinical evaluation includes blood chemistries (acute care, hepatic panel, and mineral panel) as well as measurements of pain (including allodynia, hyperalgesia, and hyperpathia), edema, autonomic dysfunction (altered skin color, temperature, or sudomotor activity) and extent of movement disorders.
Groups:
- Placebo First, Then Neurotropin: Receive Placebo 4 tabs b.i.d. for 5 weeks and then Neurotropin 4 tabs b.i.d. for 5 weeks (after at least 1 week washout period)
- Neurotropin First, Then Placebo: Receive Neurotropin 4 tabs b.i.d. for 5 weeks and then Placebo 4 tabs b.i.d. for 5 weeks (after at least 1 week washout period)
- Total: Total of all reporting groups
Arm/Group | Placebo First, Then Neurotropin | Neurotropin First, Then Placebo | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 0 | 2
  Between 18 and 65 years | 9 | 9 | 18
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.3 (13.2) | 46.5 (13.2) | 41.7 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 5 | 15
  Male | 1 | 5 | 6
Region of Enrollment [Number; unit: participants]
  United States | 11 | 10 | 21

OUTCOME MEASURES:

1. Primary Outcome: Visual Analogue Scale (VAS) of Pain Scores After Administration of Test Drugs (Placebo or Neurotropin )
Description: Assessments of pain severity by the patient using a visual analogue scale ranging from 0 to 100 (mm), with 0 = no pain and 100 = maximal pain level. When it is difficult to recruit the patients, the interim analysis using these data is performed after completion of the study of first 16 patients (target number is 30). The data from 16 patients was analyzed while investigators were blinded to the treatment code (Drug A and B) provided by the NIH pharmacy. Only after the analysis was completed was the code unblinded. Placebo or Neurotropin" in place of "drug A or drug B.
Time Frame: VAS of each patient is measured after each 5-week treatment interval with placebo or Neurotropin.
Measure: Mean (Standard Error); unit: mm
Groups:
- VAS After Placebo Treatment First in G-1: This group received placebo 4 tabs b.i.d. for 5 weeks first. VAS was determined at the end of the 5 week-treatment.
- VAS After Neurotropin Treatment Second in G-1: This group received Neurotropin 4 tabs b.i.d. for 5 weeks after at least 1 week "washout" period following the first 5 week interval on placebo. VAS was determined at the end of the 5 week-treatment of Neurotropin.
- VAS After Neurotropin Treatment First in G-2: This group received Neurotropin 4 tabs b.i.d. for 5 weeks first. VAS was determined at the end of the 5 week-treatment.
- VAS After Placebo Treatment Second in G-2: This group received placebo 4 tabs b.i.d. for 5 weeks after at least 1 week "washout" period following the first 5 week interval on Neurotropin. VAS was determined at the end of the 5 week-treatment of placebo.
Arm/Group | VAS After Placebo Treatment First in G-1 | VAS After Neurotropin Treatment Second in G-1 | VAS After Neurotropin Treatment First in G-2 | VAS After Placebo Treatment Second in G-2
Number analyzed (Participants) | 7 | 7 | 9 | 9
mm | 33.6 (11.1) | 38.3 (8.8) | 36.0 (7.6) | 31.1 (7.7)
Statistical Analysis 1: Comparison: VAS After Placebo Treatment First in G-1 vs VAS After Neurotropin Treatment Second in G-1 vs VAS After Neurotropin Treatment First in G-2 vs VAS After Placebo Treatment Second in G-2; Data from 16 patients is analyzed using one-sided paired t-test without breaking treatment code (Drug A or B, without knowing which drug is Neurotropin or Placebo) to determine if (1) the study should be terminated (if 0.0058 ≤ p), (2) the study should be terminated with rejection of the null hypothesis that there are no differences between Drug A and Drug B (p ≥ 0.9), or (3) the study will be continued to obtain the total of 42 patients (0.0058 ≤ p ≤ 0.9); Test type: Superiority or Other; p = 0.0058, t-test, 1 sided

2. Primary Outcome: Numeric Rating Scale (NRS) of Pain Scores After Administration of Test Drugs (Neurotropin or Placebo)
Description: Assessments of pain severity by the patient using a numeric rating scale ranging from 0 to 10 as a verbal response where 0 = no pain and 10 =maximal pain. When it is difficult to recruit the patients, the interim analysis using these data is performed after completion of the study of first 16 patients (target number is 30). The data from 16 patients was analyzed while the investigators are blinded to the treatment code (Drug A or B) provided by the NIH pharmacy. Only after the analysis was completed was the code unblinded. Placebo or Neurotropin" in place of "drug A or drug B.
Time Frame: NRS of each patient is measured after each five-week treatment interval with placebo or Neurotropin.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- NRS After Placebo Treatment First in G-1: This group received placebo 4 tabs b.i.d. for 5 weeks first. NRS was determined at the end of the 5 week-treatment.
- NRS After Neurotropin Treatment Second in G-1: This group received Neurotropin 4 tabs b.i.d. for 5 weeks after at least 1 week "washout" period following the first 5 week interval on placebo. NRS was determined at the end of the 5 week-treatment of Neurotropin.
- NRS After Neurotropin Treatment First in G-2: This group received Neurotropin 4 tabs b.i.d. for 5 weeks first. NRS was determined at the end of the 5 week-treatment.
- NRS After Placebo Treatment Second in G-2: This group received placebo 4 tabs b.i.d. for 5 weeks after at least 1 week "washout" period following the first 5 week interval on Neurotropin. NRS was determined at the end of the 5 week-treatment of placebo.
Arm/Group | NRS After Placebo Treatment First in G-1 | NRS After Neurotropin Treatment Second in G-1 | NRS After Neurotropin Treatment First in G-2 | NRS After Placebo Treatment Second in G-2
Number analyzed (Participants) | 7 | 7 | 9 | 9
units on a scale | 3.0 (1.1) | 3.3 (0.9) | 4.0 (0.8) | 3.1 (0.8)
Statistical Analysis 1: Comparison: NRS After Placebo Treatment First in G-1 vs NRS After Neurotropin Treatment Second in G-1 vs NRS After Neurotropin Treatment First in G-2 vs NRS After Placebo Treatment Second in G-2; Data from 16 patients is analyzed using one-sided paired t-test without breaking treatment code (Drug A or B) to determine if (1) the study should be terminated (if 0.0058 ≤ p), (2) the study should be terminated with rejection of the null hypothesis that there are no differences between Drug A and Drug B (p ≥ 0.9), or (3) the study will be continued to obtain the total of 42 patients (0.0058 ≤ p ≤ 0.9); Test type: Superiority or Other; p = 0.0058, t-test, 1 sided

3. Primary Outcome: McGill Pain Questionnaire (MPQ) of Scores After Administration of Test Drugs (Neurotropin or Placebo)
Description: Assessments of pain severity by the patient using a McGill Pain Questionnaire which consists of 3 major classes of word descriptors-sensory, affective and evaluative - that are used by patients to specify subjective pain experience. Each word chosen from descriptor responses to 20 questions is given a value and the sum of the values of the responses provides a score which is an index of the pain severity with a minimum value of 20 and a maximal value of 78. When it is difficult to recruit the patients, the interim analysis using these data is performed after completion of the study of first 16 patients (target number is 30). The data from 16 patients was analyzed while investigators are blinded to the treatment code (drug A or B) provided by the NIH pharmacy. Only after the analysis was completed was the code unblinded. Placebo or Neurotropin" in place of "drug A or drug B.
Time Frame: MPQ of each patient is measured after each five-week treatment interval with drug A or drug B.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- MPQ After Placebo Treatment First in G-1: This group received placebo 4 tabs b.i.d. for 5 weeks first. MPQ was determined at the end of the 5 week-treatment.
- MPQ After Neurotropin Treatment Second in G-1: This group received Neurotropin 4 tabs b.i.d. for 5 weeks after at least 1 week "washout" period following the first 5 week interval on placebo. MPQ was determined at the end of the 5 week-treatment of Neurotropin.
- MPQ After Neurotropin Treatment First in G-2: This group received Neurotropin 4 tabs b.i.d. for 5 weeks first. MPQ was determined at the end of the 5 week-treatment.
- MPQ After Placebo Treatment Second in G-2: This group received placebo 4 tabs b.i.d. for 5 weeks after at least 1 week "washout" period following the first 5 week interval on Neurotropin. MPQ was determined at the end of the 5 week-treatment of placebo.
Arm/Group | MPQ After Placebo Treatment First in G-1 | MPQ After Neurotropin Treatment Second in G-1 | MPQ After Neurotropin Treatment First in G-2 | MPQ After Placebo Treatment Second in G-2
Number analyzed (Participants) | 7 | 7 | 9 | 9
units on a scale | 22.4 (5.9) | 33.1 (4.0) | 25.4 (4.9) | 27.1 (5.7)
Statistical Analysis 1: Comparison: MPQ After Placebo Treatment First in G-1 vs MPQ After Neurotropin Treatment Second in G-1 vs MPQ After Neurotropin Treatment First in G-2 vs MPQ After Placebo Treatment Second in G-2; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0058, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: Adverse event information will be collected during the treatments and 5 weeks after the completion of study.
Description: Advese event information will be collected by blood test, weekly questionnaire, and self-report of patients.
Arm/Group | Placebo First, Then Neurotropin | Neurotropin First, Then Placebo
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/10
Other Adverse Events (participants affected / at risk) | 1/11 | 0/10
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo First, Then Neurotropin (N=11) | Neurotropin First, Then Placebo (N=10)
worsening of pain (Nervous system disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Because of the difficulty in patient recruitment, the interim analysis was performed for the first 16 patients (target was 30). The results are inconclusive due to large variations in pain scores associated with insufficient the number of patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes